CLINICAL TRIAL: NCT03715400
Title: Mobile Virtual Positive Experiences for Anhedonia
Acronym: MVR
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Restrictions for in-person study procedures
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Mobile Virtual Reality Study
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Anhedonia; Virtual Reality; Depression; Mood Disorders; Stress; Anxiety
Keywords: Virtual Reality; Depression; Stress; Anxiety; Treatment
MeSH Terms: conditions — Anhedonia; Depression; Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will not undergo the positive virtual reality training program. Instead, they will complete all self-report and behavioral measures and have the option to experience the positive virtual reality training program upon the conclusion of the study.
- Positive Virtual Reality Training Intervention (Experimental): The experimental group will undergo the positive virtual reality training program, which consists of 7 virtual reality (VR) sessions to be completed at home after orientation to the program, in addition to all self-report and behavioral measures.
  Interventions: Behavioral: Positive Virtual Reality Training

INTERVENTIONS:
Behavioral: Positive Virtual Reality Training — Participants will undergo 7 45 minute sessions of positive virtual reality training over the course of four weeks. All assessments will be completed online at home following initial orientation to the program.
  Other Names: Mobile Virtual Reality Training
  Arms: Positive Virtual Reality Training Intervention

SUMMARY:
Anhedonia is a symptom dimension that characterizes many individuals suffering from depression, as well as some types of anxiety, psychosis, and substance use. For the most part, treatments are effective in decreasing negative affect but ineffective in improving anhedonia, with some antidepressant medications even worsening symptoms of anhedonia. Yet anhedonia is a significant marker of poor prognosis as well as suicidal ideation and actual suicide. The development of effective treatments for anhedonia is thus of paramount importance. Advances in neuroscience indicate specific targets that may underlie anhedonia that can be shifted through behavioral training. The investigators have developed such a program and found it to be effective in raising positive affect, especially for depressed or anxious individuals with anhedonia at baseline. To date, this program has been implemented by highly trained clinicians, which have supervised its implementation on a large scale. Moreover, the behavior program is dependent on readily available rewarding experiences, which anhedonia obviously challenges. Furthermore, mechanistic evaluation is impeded by intra¬- and inter-¬individual variability in exposure to rewarding stimuli. Virtual Reality (VR) offsets these barriers by repeated controlled immersion in experiences designed to enhance approach motivation, initial responsiveness to reward attainment, and reward learning. In this current study, the investigators aim to measure clinical outcomes using Virtual Reality-Reward Training (VR-RT).

DETAILED DESCRIPTION:
Anhedonia is a symptoms dimension that characterizes many individuals suffering from depression, as well as some types of anxiety, psychosis, and substance use. Anhedonia refers to deficits in positive affect as observed through 1) loss of enjoyment in pleasurable activities and/or 2) loss of desire to engage in pleasurable activities. Within depression, anhedonia is more strongly associated with the core disturbance of depressions (e.g. lassitude) than with the nonspecific symptoms that are shared without emotion disorders (e.g. insomnia). Approximately one¬-third of depressed individuals have clinically significant anhedonia symptoms, as defined by cutoffs on scales that measure enjoyment of social and physical pleasure. Anhedonia extends beyond major depression to social anxiety disorder and generalized anxiety disorder, although with a smaller magnitude of effect than depression. Anhedonia is also relevant to schizophrenia and substance use disorder. Thus, anhedonia represents a dimension of psychopathology that crosses diagnostic boundaries.

Anhedonia is associated with several indices of psychopathology. First, self¬-reported anhedonia (lower levels of positive emotion) is a robust predictor of poorer longitudinal course of symptoms of major depression across a number of prospective studies. Relatedly, the trait variance component of low positive affect prospectively predicts the onset of not only major depression, but also social anxiety disorder and generalized anxiety disorder, albeit through correlates with neuroticism. Second, anhedonia within major depression is a major predictor of suicide, and the predictive effects upon suicidal ideation persist even when controlling for other cognitive and affective symptoms of depression. Third, anhedonia is a predictor of poorer response to pharmacological treatments for depression. Some preliminary data from our laboratory replicate this relationship in terms of psychological treatments, at least for social anxiety disorder: in a sample of 75, the investigators found that low positive affect again significantly predicted poorer outcomes (b = ¬-.70, B = -¬.25, p < .05).

Approach Motivation: Dopaminergic signaling is related to the motivation for reward. In humans, neural regions most strongly linked to the approach motivation for reward include the ventral tegmental area, amygdala, and striatum, all of which are innervated by or project to dopaminergic nuclei. Phasic bursts in dopaminergic neurons in the ventral tegmental area have been shown to co¬-occur in response to violations in reward expectancy. Dopamine signaling in the nucleus accumbens (which has dense dopaminergic projections from the ventral tegmental area) is also associated with reward motivation in rodents. Increased mPFC activation may function to reduce striatal response and behavioral drive for rewarding dopaminergic stimulation. Approach motivation is also tied to reward learning, which involves Pavlovian or instrumental associations and predictions about future rewards based on past experiences. As with the approach motivation for reward, learning of reward is associated with dopaminergic signaling. Various areas of the prefrontal cortex have been implicated in decision making and reward learning, and animal research highlights areas such as the ACC, orbitofrontal cortex, vmPFC and dlPFC. Not only do depressed individuals show reduced activation in reward circuitries in anticipation of reward but reduced ventral striatum responsivity to incentive stimuli is particularly related to anhedonic symptoms. Further evidence is derived from behavioral indices in which trait anhedonia among healthy individuals correlates with choosing easy tasks for a small reward over harder tasks for larger rewards, indicative of less motivation (i.e., expenditure of effort) to gain reward. Also, depressed individuals make fewer higher reward/high effort choices than healthy controls, and importantly, the motivational effort they expend to obtain rewards correlates negatively with anhedonia. In self-¬report measures, dysphoric individuals expect to feel less positive emotion in future positive events and report less positive emotion in anticipation of a monetary reward compared to healthy controls, although the evidence is not entirely robust.

Responsiveness to Reward Attainment: Responsiveness to reward attainment (or hedonic capacity) is more strongly related to opioid and endocannabinoid pathways. Neural regions most strongly linked with liking of reward include the ventral striatum (representing overlap with the approach motivation component) and orbitofrontal cortex. Depressed individuals show ventral striatum hypo-activity to positive stimuli, and the hypo-activity is particularly strongly associated with symptoms of anhedonia. Furthermore, Wacker et al. (2009) established that the effects were specific to anhedonia above and beyond negative symptoms of anxiety and depression. Further evidence for deficits in initial responsiveness to attainment derives from cognitive measures, with depressed individuals showing less attention to positive stimuli than controls as measured by response latency times in dot probe tasks and eye tracking. Moreover, attention to positive information is associated with positive affect. The evidence for deficits in self-¬rated liking of reward in depressed individuals is mixed. Importantly, lower levels of self¬-reported positive emotions to positive stimuli (e.g. sweet taste test) are more strong related to anhedonia than depression.

Targeted Treatment for Anhedonia: In light of the evidence summarized above, a treatment that specifically targets reward approach motivation and learning, and responsiveness to reward attainment may be particularly potent for anhedonia. As noted, existing psychological treatments mostly target negative affect, and while behavioral activation is designed to increase engagement in pleasant activities, little attention has been given to date to how to optimize positive emotions during the planning and conduct of such activities. Drawing from affective neuroscience and experimental psychopathology, the investigators have developed a treatment that specifically targets these components of the reward system. The treatment is comprised of therapeutic techniques that directly target one or more of these subdomains. The first phase of treatment (sessions 1-7) involves modified behavioral activation (called behavioral training), which combines planning for engagement in pleasurable activities (reward approach and motivation) and reinforcement via positive mood inducing effects (reward learning) with 'in¬-the-¬moment' recounting designed to savor pleasurable moments and enhance hedonic impact (responsiveness). The second phase of treatment (sessions 8¬-13) adds two additional components to ongoing behavioral training: cognitive training designed to shift attention towards positive stimuli in the environment (reward approach motivation), reinforce associations between responses and positive outcomes (reward learning) and train motivation for positive events and emotions through imagery (reward approach motivation); and compassion training that focuses on motivating toward (reward approach motivation) and savoring positive experiences (responsiveness). The investigators found that this treatment is effective in both reducing negative affect (depression and anxiety) and improving positive affect, especially for individuals who are most anhedonic at baseline. Specifically, patients who meet entry criteria of elevated levels of depression, anxiety (somatic), or stress (worry) on the Depression, Anxiety and Stress Scale (DASS-21), and who are at least moderately impaired according to the Sheehan Disability Scale (SDS), are randomly assigned to receive treatments aimed at increasing reward sensitivity (Positive Affect Treatment, PAT) or at reducing threat sensitivity (Negative Affect Treatment, NAT). Here the investigators present data from the first 61 enrolled patients (N=20 PAT and N=41 NAT) who began the 15 ¬treatment session protocol. Self-¬reported symptoms of depression (DASS-¬D) and stress (DASS-¬S) decreased from a severe range at pre-¬treatment to a normal range at post-¬treatment in PAT and NAT (DASS¬-D: Cohen's d=1.89 and 1.41, respectively; DASS¬-S: d=1.35 and d=1.65, respectively). Self¬-reported anxiety (DASS¬-A) decreased from extremely severe to normal for PAT and from moderate to mild for NAT (d=1.02 and 1.47). The investigators found significant improvements for our anhedonia outcome measure, Positive and Negative Affect Schedule Positive Scale (PANAS-¬P). Positive affect improved linearly in both treatment, but significantly greater changes occurred with PAT (d=1.40) versus NAT (d=.59) (Group x Time; p=.001). Only PAT significantly and satisfactorily normalized deficits in positive affect (changes from 20th to 46th percentile on the scale developed by Crawford Henry, 2004. In NAT treatment, levels of PANAS-¬P remained lower than the population average (change from 18th to 32nd percentile).

Virtual Reality-Reward Training: While our "reward training" treatment has a strong preliminary efficacy signal, it is dependent on delivery by highly trained clinicians, which reduces its scalability and accessibility to large section of the population. Furthermore, evaluation of mechanisms is somewhat impeded by variability both within the between individuals in terms of rate of exposure to rewarding stimuli. Finally, chronically anhedonic individuals, especially those with limited social contact and therefore lack of social reinforcement, may be faced with difficulties when asked to repeatedly engage in rewarding experiences. Repeated imagining of positive outcomes from multiple scenarios has already been shown to be an effective means for raising positive affect. However, imagery alone provides limited control over the content of images and is dependent upon an individual's ability to imagine vividly. Virtual reality provides a vehicle for repeated programmatic immersion in rewarding experiences that can include training to identify positive stimuli, sustain attention upon positive stimuli, receive reinforcement for such attention, and notice mood enhancing effects, with training extending from primary reward (e.g. physical and social) to acts of generosity/loving kindness. This type of automated training offers the potential to eventually become a self-¬guided treatment which would increase implementation on a large scale. Furthermore, it offers a mechanistic dose-¬response evaluation since the dosage of rewarding experiences within virtual reality can be fully controlled. Virtual reality with relaxing scenes has been shown to increase ratings of happiness. Virtual reality has already been tested and shown to be an effective tool for raising positive affect in patients with chronic or terminal medical conditions.

Potential participants will complete a brief online screener to verify eligibility. Eligible participants will be randomized to VR-RT or a delayed waitlist control condition. All participants will complete a Baseline assessment at Week 0 through Qualtrics that measures symptoms of anhedonia, depression, and anxiety. Participants randomized to VR-RT will be provided with VR viewers to allow them to use their smartphone devices to view virtual reality scenes.

Participants will have the option to proceed with online screening through this webpage, which will initiate the pre-screening process. During pre-screening, participants will be asked to answer a brief screener. If participants are eligible after this step, they will continue with prescreening by completing the 1) BAS, 2) DASS-21, and 3) SDS. Participants will be eligible based on meeting the following dimensional score cutoffs: BAS (Reward Drive subscale score of ≤ 11, Reward Sensitivity Subscale score of ≤ 11, or Responsiveness subscale score of ≤ 16), DASS-21 score above mild/moderate in any subscale, and SDS score of ≥6. Those who meet the appropriate score cutoffs listed above will be redirected to the study information sheet and online consent form. On the online consent form, participants will be asked to 1) agree to participate in the study, 2) confirm willingness to be contacted for future studies, and 3) confirm willingness to share data with other investigators. After providing online consent, participants will provide contact information (which will include phone verification and email verification steps), age and sex, and preferred mode of contact through a secured registration system. Once this information is collected, participants will receive a notification that they will be contacted within three business days to complete the final screening step by phone. If participants are not eligible after completing the online screening or decline to provide consent, they will be sent a notification of their ineligibility and a list of resources. If the participants are found eligible, they will be randomized to the treatment or waitlist control group and scheduled for all of the VR-¬RT sessions and assessments.

At each assessment, the participant will complete the PANAS-SF (at beginning and end), MASQ-AD 14 item, DASS-21, Ruminative Responses Scale, SDS, EEfRT task, and Pizzagalli task. Each of these sessions is expected to take approximately one hour, with the exception of the Treatment condition Baseline, which will take roughly 2.5 hours, as it includes an initial orientation to the VR program, they will be instructed how to access the VR scenes online and view them using the virtual reality viewer, as well as how to use Qualtrics to guide their recall of the VR scenes and autobiographical memories. Please see the attached document "Amended Participant Timeline" for a Participant timeline.

Description of Virtual Reality Reward Training (VR-RT): VR-RT will be scheduled twice weekly for with each lasting roughly 45 minutes (7 sessions, 4 weeks total). These sessions will occur at a comfortable, private location (e.g. at home) with a sufficiently strong Wi-Fi connection chosen at the participant's discretion. We have determined that UCLA's campus has sufficiently strong Wi-Fi connection to complete the VR-RT viewings and tasks. Participants will therefore be offered the option to complete their sessions on campus in the laboratory of Dr. Craske in the Life Sciences Building.

The first session will consist of an overview of the treatment, instruction in the use of the virtual reality equipment, and Session 1 of VR-RT. Each session will involve unique virtual reality scenes. All virtual reality scenes will contain physical (e.g. walking through a beautiful forest) and/or social (e.g. being welcomed as entering a social gathering) reward-related sub-scenes in which higher-intensity rewarding stimuli are embedded and are to be discovered through searching (e.g. sun filtering through the forest in one of several hiking trials; being invited to join a group within a larger social gathering); negative sub-scenes may also be embedded (e.g. clouds looming overhead; a group who ignore the participant) in order to emphasize focus on the positive aspects of the scenes. Some of the social reward scenes will involve acts of generosity and loving kindness.

Each session will be comprised of three components: 1) Preparation. Participants will be given a description of the virtual scene to which they will be exposed. They will be informed that their task is to become as fully immersed in the scene as possible, to notice their emotions, physical reactions and thoughts as they participate, and to move away from embedded negative stimuli and discover embedded higher intensity rewarding stimuli through searching behavior and to move away from embedded negative scenes; this represents training in goal setting and approach motivation. Participants will rate their mood using the International Positive and Negative Affective Schedule Short Form (I-PANAS-SF) to assess positive affect and negative affect, anchored to current mood states. They will then connect their smartphone to the virtual reality equipment, queuing up the VR video for that session. 2) Experience. Each session will consist of two to six videos and average approximately 15 minutes. 3) Evaluate and Recount. Participants will complete a Post- VR I-PANAS-SF. Participants will type into Qualtrics their recollection of the VR scene(s). They will then listen to a guided mindfulness summary of the scene(s) they just watched. Participants will then type into Qualtrics their recollection of an autobiographical memory; the autobiographical memory they recall will be prompted by the program, differing by session. Participants will then listen to a guided mindfulness recording that prompts them to recall their own, prompted autobiographical memory. In doing so, the training targets savoring or attainment of reward and reward learning (i.e., my mood is changed by this activity). Participants will then rate their mood again according to the I-PANAS-SF.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English
* below the population mean on either the Behavioral Activation Scale (BAS) Reward Drive subscale (score of ≤ 11), or BAS Responsiveness subscale (score of ≤16)
* score in mild-moderate range on DASS-21 following established score cutoffs: Depression (10-27); at least a score of Anxiety (8-14); and a score of at least Stress (15-25)
* Sheehan Disability Scale (SDS) overall score must be ≥ 6
* agree to refrain from initiating other psychosocial treatments throughout the duration of the study

Exclusion Criteria:

* Lifetime history of bipolar disorder, psychosis, intellectual disabilities, or organic brain damage
* substance use disorder in the past 6 months
* current use of psychotropic medications
* currently pregnant or planning to become pregnant
* self-reported frequent motion sickness, self-reported seizures within the last year and/or a diagnosis of epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in anhedonia | Baseline to Post-treatment (4 weeks)
  Change in anhedonia as measured by the anhedonia subscale of the Mood and Anxiety Symptom Questionnaire (MASQ) (max: 110, min: 22, with a higher score indicating higher anhedonia)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Craske, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No